CLINICAL TRIAL: NCT07175116
Title: Use of Advanced Fixation Dressings in Reducing Central Venous Catheter-related Bloodstream Infections in a Paediatric Intensive Care Unit
Brief Title: Advanced Dressings for CVC Infection Prevention in PICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Collaborators: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, MANUEL PABON CARRASCO, Principal Investigator, Faculty of Nursing, Physiotherapy and Podiatry, University of Seville, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: US-PICU-CV
Record Dates: First submitted 2025-09-05; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Catheter-Related Infections; Central Venous Catheters; Bloodstream Infection; Pediatric Intensive Care Units
MeSH Terms: conditions — Catheter-Related Infections; Sepsis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This was a single-blind trial. The outcomes assessor was blinded to group allocation. Participants and care providers were aware of the dressing used
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental - Chlorhexidine gluconate-impregnated dressing (Experimental): Participants receive advanced transparent dressings impregnated with chlorhexidine gluconate at the CVC insertion site.
  Interventions: Device: 3M™ Tegaderm™ Antimicrobial Transparent Dressing (chlorhexidine gluconate-impregnated)
- Control - Conventional transparent dressing (Active Comparator): Participants receive standard transparent polyurethane dressing without antimicrobial activity at the CVC insertion site.
  Interventions: Device: Conventional transparent polyurethane dressing

INTERVENTIONS:
Device: 3M™ Tegaderm™ Antimicrobial Transparent Dressing (chlorhexidine gluconate-impregnated) — Individually applied transparent dressing containing chlorhexidine gluconate (0.5-1 mg/cm²) for antimicrobial protection at the central venous catheter insertion site. The dressing maintains site visibility, reduces catheter manipulation frequency, and provides sustained release of chlorhexidine to lower colonisation and bloodstream infection risk.
  Arms: Experimental - Chlorhexidine gluconate-impregnated dressing
Device: Conventional transparent polyurethane dressing — Transparent polyurethane dressing without antimicrobial impregnation, applied at the central venous catheter insertion site. This dressing allows site inspection and is widely used in standard paediatric intensive care protocols but provides no antimicrobial activity.
  Arms: Control - Conventional transparent dressing

SUMMARY:
Randomised, single-blind clinical trial comparing chlorhexidine gluconate-impregnated transparent dressings versus conventional transparent dressings in the prevention of central venous catheter-related bloodstream infections (CVC-BSI) in paediatric patients admitted to a tertiary hospital PICU. Outcomes include incidence of BRCVC, catheter colonisation, dressing-related skin complications, and number of dressing changes.

ELIGIBILITY:
Inclusion Criteria:

* Admission to paediatric intensive care unit (PICU)
* Central venous catheter placement (central or peripherally inserted)
* Informed consent obtained from parent/legal guardian

Exclusion Criteria:

* Known immunological disorders
* Neutropenia (<500/mm³)
* Pre-existing colonisation or infection with multidrug-resistant organisms

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of central venous catheter-related bloodstream infection (CVC-BSI) | Baseline to 4 weeks or until catheter removal
  CVC-BSI confirmed by clinical signs and positive blood culture according to Bacteriemia Zero protocol.

SECONDARY OUTCOMES:
Catheter colonisation rate | At catheter removal (up to 14 days after insertion)
  Positive culture of catheter tip (>15 CFU/mL) according to standard microbiological protocol.
Skin complications at insertion site | Up to 4 weeks
  Erythema, pruritus or dermatitis at the catheter insertion site documented by clinical observation.
Number of dressing changes per patient | Up to 4 weeks
  Total number of dressing replacements per patient recorded during catheterisation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen del Rocío - Hospital Infantil, Seville, Sevilla, Spain

IPD SHARING:
Plan to Share IPD: Undecided